CLINICAL TRIAL: NCT00795054
Title: The Financial Impact of Allogeneic Stem Cell Transplantation on Patient and Family: A Pilot Study
Brief Title: The Financial Impact of Allogeneic Stem Cell Transplantation on Patient and Family
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: CIBMTR HS 07-02
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Financial Impact of Stem Cell Transplantation
Keywords: Stem cell transplantation; Financial impact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- allogeneic stem cell recipients: Pediatric and adult allogeneic stem cell transplant recipients and their care givers.
  Interventions: Other: Household financial data collection

INTERVENTIONS:
Other: Household financial data collection — Baseline financial survey pre-transplant, financial diary post-transplant every two weeks for 3 months, and financial questionnaire via phone survey at 6, 12, 18 and 24 months post-transplant.

SUMMARY:
The purpose of this pilot study is to determine the feasibility of conducting a study of out-of-pocket costs and the long-term financial impact of allogeneic stem cell transplant.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) is the indicated treatment for many life-threatening illnesses affecting both adults and children. Transplant recovery and late effects require long-term medical care. At the same time that the family faces a medical crisis, a resulting financial crisis may also be pending, but is often pushed to the background due to the necessity of first preserving life. A large proportion of patients undergoing HSCT incur significant financial burden from out-of-pocket costs and a decrease in household income. Predetermined variables, both medical and demographic, gathered at the pre-transplant clinical consultation have the potential to predict the patients at greatest financial risk. This study will describe both the out-of-pocket costs and the income changes that may result from HSCT to help patients and their caregivers have a clearer picture of these costs and develop a financial plan. Health care providers can utilize this information to better inform patients and connect them to resources.

ELIGIBILITY:
Inclusion Criteria:

1. Adult recipients and parents/guardians of pediatric (age 0-17 years) recipients of allogeneic HSCT
2. Recipient has a primary caregiver, who is a member of the recipient's household
3. Allogeneic HSCT using any donor cell source (related, unrelated, or cord blood)
4. Any age at HSCT
5. Diagnosis of primary disease for which HSCT is being performed must have been made within two years prior to transplantation
6. Adult recipients, parents/guardians of pediatric recipients, and primary caregivers should be able to read, write, and understand the English language
7. Signed informed consent from adult patient, caregiver and/or parent/guardian for study participation
8. Signed consent to participate in the Center for International Blood and Marrow Transplant Research (CIBMTR) research database.

Exclusion Criteria:

1. Recipients who have had a previous HSCT (autologous or allogeneic)
2. Households with more than one transplant recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult allogeneic stem cell transplant recipients and their care givers from three U.S. transplant medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To study the feasibility of using a patient maintained diary to capture out-of-pocket costs over the first 3 months following allogeneic HSCT | Pre-transplant and for 3 months post-transplant

SECONDARY OUTCOMES:
To determine the feasibility of conducting interviews to collect financial information at 6, 12, 18 and 24 months after allogeneic HSCT | 6, 12, 18 and 24 month time points post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Navneet Majhail, MD, MS, Study Chair — University of Minnesota / CIBMTR; Douglas Rizzo, MD, MS, Study Chair — Medical College of Wisconsin / CIBMTR
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Medical College of Wisconsin, Milwaukee, Wisconsin